CLINICAL TRIAL: NCT04763408
Title: A Multicentre, Observational, Phase 4 Study to Evaluate the Safety and Tolerability of Lenvatinib in Patients With Advanced or Unresectable Hepatocellular Carcinoma (STELLAR)
Brief Title: A Study to Evaluate the Safety and Tolerability of Lenvatinib in Participants With Advanced or Unresectable Hepatocellular Carcinoma
Acronym: STELLAR
Status: Completed | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E7080-M000-508
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Lenvatinib; Advanced or unresectable carcinoma hepatocellular; E7080
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lenvatinib: Participants with advanced or unresectable HCC will initiate treatment with lenvatinib capsules based on physicians decision and will be observed until withdrawal of consent, loss to follow-up, death or until the end of the study (up to 7 years) whichever occurs first.
  Interventions: Drug: Lenvatinib
- Sorafenib: Participants with advanced or unresectable HCC will initiate treatment with sorafenib tablets based on physicians decision and will be observed until withdrawal of consent, loss to follow-up, death or until the end of the study (up to 7 years) whichever occurs first.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Lenvatinib — Oral capsules.
  Other Names: Lenvima; E7080
  Groups: Lenvatinib
Drug: Sorafenib — Oral tablets.
  Groups: Sorafenib

SUMMARY:
The primary purpose of this study is to further characterise the hepatotoxicity in participants with advanced or unresectable hepatocellular carcinoma (HCC) treated with lenvatinib, and to further characterise the overall safety profile (serious adverse events [SAEs], grade 3 to 5 adverse events [AEs], dose modifications and discontinuations due to AEs) in participants with advanced or unresectable HCC treated with lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with advanced or unresectable HCC for whom a decision has been made by the treating physician (at their discretion) to initiate lenvatinib or sorafenib treatment, within the prescribing conditions of the approved product label
2. Participants must provide signed informed consent to participate in the study within 31 days of initiating treatment with lenvatinib or sorafenib

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participant with advanced or unresectable hepatocellular carcinoma.
Sampling Method: Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Hepatotoxicity Treatment-emergent Adverse Events (TEAEs) With Lenvatinib | Up to 7 years
Number of Participants With SAEs With Lenvatinib | Up to 7 years
Number of Participants With Grade 3 to 5 AEs With Lenvatinib | Up to 7 years
  AEs are defined as undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment with lenvatinib. AEs will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE). Here Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activity of daily living, Grade 4: life-threatening consequences; urgent intervention indicated and Grade 5: death related to AEs.
Number of Participants with one or More TEAEs Leading to Dose Modifications and Treatment Discontinuations of Lenvatinib | Up to 7 years
  Number of participants with one or more TEAEs Leading to Dose Modifications and Treatment Discontinuations of Lenvatinib will be collected at the discretion of the treating physician and in accordance with the prescribing information.

SECONDARY OUTCOMES:
Duration of Lenvatinib and Sorafenib Treatment | Up to 7 years
Number of Participants With Dose Interruption and Dose Reduction for Lenvatinib | Up to 7 years
Relative Dose Intensity of Lenvatinib and Sorafenib | Up to 7 years
  Relative Dose Intensity is defined as the amount of drug administered divided by the total dose specified by the corresponding standard regimen.
Overall Survival (OS) For Lenvatinib and Sorafenib | Up to 7 years
  OS is defined as the time from the start of lenvatinib and sorafenib treatment to date of death from any cause.
Number of Participants With Dose Interruption and Dose Reduction for Sorafenib | Up to 7 years
Number of Participants With Hepatotoxicity TEAEs With Sorafenib | Up to 7 years
Number of Participants With SAEs With Sorafenib | Up to 7 years
Number of Participants With Grade 3 to 5 AEs With Sorafenib | Up to 7 years
  AEs are defined as undesirable events not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment with sorafenib. AEs will be graded using NCI CTCAE. Here Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activity of daily living, Grade 4: life-threatening consequences; urgent intervention indicated and Grade 5: death related to AEs.
Number of Participants with one or More TEAEs Leading to Dose Modifications and Treatment Discontinuations of Sorafenib | Up to 7 years
  Number of participants with one or more TEAEs Leading to Dose Modifications and Treatment Discontinuations of Sorafenib will be collected at the discretion of the treating physician and in accordance with the prescribing information.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (3):
  - California Liver Research Institute, Pasadena, California
  - Montefiore Medical Center, The Bronx, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Monash Health, Monash Medical Centre, Clayton, Victoria
- Austria (4):
  - Universitätsklinikum Innsbruck, Innsbruck, Tyrol
  - Klinikum Klagenfurt Am Woerthersee, Klagenfurt
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
- Germany (5):
  - Eisai Trial Site #3, Cologne, North Rhine-Westphalia
  - Eisai Trial Site #5, Mainz, Rhineland-Palatinate
  - Eisai Trial Site #2, Berlin
  - Eisai Trial Site #6, Munich
  - Eisai Trial Site #1, Ulm
- Italy (6):
  - Ospedale del Mare, Napoli, Campania
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli, Rome, Lazio
  - Azienda Ospedaliero Universitaria Di Cagliari, Monserrato Cagliari, Sardinia
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna
- Portugal (4):
  - Hospital Garcia de Orta, Almada, Setúbal District
  - Instituto Português de Oncologia Francisco Gentil Centro Regional de Oncologia de Coimbra EPE, Coimbra
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Trás Os Montes E Alto Douro EPE, Vila Real
- Budgetary Institution of the Chuvash Republic-The Republican Clinical Oncologic Dispensary-Cheboksar, Cheboksary, Chuvashskaya Respublika, Russia
- Spain (13):
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Virgen de La Arrixaca, El Palmar, Murcia
  - Hospital General Universitario de Alicante, Alicante
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - CHUS - H. Clinico U. de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Karolinska Universitetssjukhuset Huddinge, Stockholm, Sweden
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Barts Health NHS Trust - Charterhouse Square, London
  - Royal Free London NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.